CLINICAL TRIAL: NCT06775431
Title: Comparison of Prophylactic Intravenous Pethidine Versus Intrathecal Pethidine in Preventing Post Spinal Shivering in Caesarean Section
Brief Title: Comparing Prophylactic Intravenous Pethidine and Intrathecal Pethidine in Preventing Post Spinal Shivering in Caesarean Section
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0306931
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Pregnant Women
Keywords: post spinal shivering; IV pethidine; intrathecal pethidine; caesarean section
MeSH Terms: interventions — Meperidine; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVGroup (Active Comparator): This group will receive IV 0.5mg/kg Pethidine as premedication mixed into 10 ml normal saline slowly IV
  Interventions: Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection
- Intrathecal Group (Active Comparator): This group will receive intrathecal Pethidine 0.2 mg/kg and 2.5 ml Bupivacaine 0.5%
  Interventions: Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection administered intrathecally

INTERVENTIONS:
Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection — Pethidine will be administered intravenously in group A 0.5 mg/kg as premedication
  Arms: IVGroup
Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection administered intrathecally — 0.2 mg/kg pethidine in trathecally will be administered with bupivacaine 0.5% in group B
  Arms: Intrathecal Group

SUMMARY:
The goal of this clinical trial is to assess the effect of IV pethidine and intrathecal pethidine on the incidence, onset, duration, and intensity of shivering in females undergoing caesarean section. The main question it aims to answer is: which route is more efficacious in preventing shivering.

Researchers will compare IV pethidine and intrathecal pethidine to see their effects on post spinal shivering, their effects on hemodynamic stability, nausea, vomiting, and sedation.

DETAILED DESCRIPTION:
This study will be a single blinded, randomized, prospective controlled study. After obtaining written informed consents, 86 patients of American Society of Anesthesiologists physical status II, aged 20-40 years old, undergoing spinal anesthesia for elective cesarean section will be investigated at El-Shatby University Hospital.

The patients will be randomized into two groups of n=43 each using a computer-generated sequence. Allocation concealment will be done using sealed envelope technique. Depending on the group allocation either to receive IV Pethidine 0.5mg/kg (Group A n=43 patients) as premedication mixed into 10 ml isotonic saline slowly IV or intrathecal Pethidine 0.2 mg/kg and 2.5 ml Bupivacaine 0.5% (Group B n=43 patients). SA will be given at either L3-L4 or L4-L5 in the sitting position by the anesthetist using 22-25-gauge Quincke spinal needles. Patients will be covered with drapes but not actively warmed. 10mg ephedrine will be given if the patient becomes hypotensive (hypotension is defined as a decrease in MAP of >20% from the baseline). 0.5 mg atropine IV will be given if HR less than 50 beats/min. Rescue 4 mg ondansetron IV will be given for vomiting episodes. Room temperature will be maintained about 21 - 24ºC during the perioperative period in the OR and in the PACU, using temperature control system. The presence of shivering will be observed and graded after spinal injection by using Tsai and Chu Scale.

The following parameters will be measured:

1. Vital signs (heart rate, and blood pressure) will be measured at baseline and every 5 minutes after administration of the drug for 30 minutes, then every 15 minutes till the end of surgery and every 30 minutes in the first two hours postoperatively
2. Body temperature (in degrees Celsius), will be measured, using axillary thermometer before drug administration then every 15 minutes till the end of surgery. After surgery, axillary temperature will be measured every 30 minutes for 2 hours.
3. Using Tsai and Chu Scale for shivering assessment, the incidence, duration, time interval from onset of spinal block to shivering occurrence, and intensity of shivering will be recorded every 15 minutes during the surgery and every 30 minutes for 2 hours postoperatively in the recovery room.
4. Complications of the drugs, such as nausea, vomiting and sedation will be recorded.

The primary aim of this study will be to assess the effect of IV pethidine and intrathecal pethidine on the incidence, onset, duration, and intensity of shivering. The secondary aims will be to assess the effect of different routes of administration of the drug on hemodynamic stability, nausea, vomiting, and sedation.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

1. contraindications to spinal
2. uncontrolled hypertension, diabetes mellitus, hepatic, pulmonary diseases, and thyroid disease
3. obesity (BMI >35)
4. drug allergy
5. temperature below 36 degrees celcius or above 37.5 degrees celcius

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females undergoing caesarean section
Enrollment: 86 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Shivering incidence | every 15 minutes during the surgery and every 30 minutes for 2 hours postoperatively
  The primary aim of this study will be to assess the effect of IV pethidine and intrathecal pethidine on the incidence of shivering
Onset of shivering | every 15 minutes during the surgery and every 30 minutes for 2 hours postoperatively
  The primary aim of this study will be to assess the effect of IV pethidine and intrathecal pethidine on the onset of shivering
Duration of shivering | every 15 minutes during the surgery and every 30 minutes for 2 hours postoperatively
  The primary aim of this study will be to assess the effect of IV pethidine and intrathecal pethidine on the duration of shivering
Shivering intensity | every 15 minutes during the surgery and every 30 minutes for 2 hours postoperatively
  The primary aim of this study will be to assess the effect of IV pethidine and intrathecal pethidine on the intensity of shivering, using the Tsai and Chu Scale
  The intensity of shivering using Tsai and Chu scale is measured as follows:
  0: no shivering
  1. piloerection or peripheral vasoconstriction, but no visible shivering
  2. muscular activity in only one muscle group
  3. muscular activity in more than one muscle group, but not generalized
  4. shivering involving the whole body

SECONDARY OUTCOMES:
Hemodynamic stability | at baseline and every 5 minutes after administration of the drug for 30 minutes, then every 15 minutes till the end of surgery and every 30 minutes in the first 2 hours postoperatively
  The secondary outcome is to assess the effect of different routes of administration of the drug on hemodynamic stability, by measuring the heart rate and blood pressure
Incidence of vomiting | from administration of spinal till 2 hours postoperatively
  The secondary outcome is to assess the effect of different routes of administration of the drug on incidence of vomiting
Incidence of sedation | from administration of spinal till 2 hours postoperatively
  The secondary outcome is to assess the effect of different routes of administration of the drug on incidence of sedation

OTHER OUTCOMES:
Body Temperature | before administration of the drug, then every 15 minutes till the end of surgery and every 30 minutes for 2 hours postoperatively
  Body temperature will be measured using an axillary thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- El-Shatby University Hospital, Alexandria, Alexandria Governorate, Egypt